CLINICAL TRIAL: NCT03292653
Title: An Exploratory, Randomized, Double-blind, Placebo-controlled, Parallel Arm Trial of the Safety and Pharmacodynamic Activity of Sotagliflozin in Hemodynamically Stable Patients Hospitalized With Worsening Heart Failure
Brief Title: Safety, Tolerability and Pharmacodynamic Activity of Sotagliflozin in Hemodynamically Stable Participants With Worsening Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 1st two cohorts provided the required data, therefore 3rd cohort was not deemed necessary
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDY15079; 2017-002774-39 (EudraCT Number); U1111-1190-7962 (Other: UTN)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Cardiac Failure Aggravated
MeSH Terms: interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants were randomized to matching placebo to sotagliflozin administered as two tablets, once daily, before the first meal of the day in the double-blind treatment period for up to 14 days.
  Interventions: Drug: Placebo
- Sotagliflozin 200 mg (Experimental): Participants were randomized to Sotagliflozin 200 mg administered as 1 sotagliflozin tablet and 1 matching placebo tablet, once daily, before the first meal of the day in the double-blind treatment period for up to 14 days.
  Interventions: Drug: Sotagliflozin; Drug: Placebo
- Sotagliflozin 400 mg (Experimental): Participants were randomized to Sotagliflozin 400 mg administered as two 200 mg sotagliflozin tablets, once daily, before the first meal of the day in the double-blind treatment period for up to 14 days.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Sotagliflozin — Pharmaceutical form: Tablet; Route of administration: Oral
  Other Names: SAR439954
  Arms: Sotagliflozin 200 mg; Sotagliflozin 400 mg
Drug: Placebo — Pharmaceutical form: Tablet; Route of administration: Oral
  Arms: Placebo; Sotagliflozin 200 mg

SUMMARY:
Primary Objectives:

* Assess the safety and tolerability of sotagliflozin in hemodynamically stable participants with worsening of heart failure, compared to placebo.
* Estimate the effects of sotagliflozin on plasma volume changes in hemodynamically stable participants with worsening of heart failure, compared to placebo.

Secondary Objectives:

* Explore the effect of sotagliflozin on erythropoiesis, as assessed by changes in plasma erythropoietin levels, in hemodynamically stable participants with worsening of heart failure, compared to placebo.
* Explore the effect of sotagliflozin on changes in plasma N-terminal prohormone of brain natriuretic peptide (NT-proBNP) levels, in hemodynamically stable participants with worsening of heart failure, compared to placebo.

DETAILED DESCRIPTION:
The total study duration will be approximately 27-40 days, including a screening period of 1-10 days, a treatment period of 14 days, and a follow-up period of 14±2 days.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent.
* 18 years of age or older.
* Participants admitted to the hospital or had urgent visit to emergency department or heart failure unit/clinic or infusion center for Congestive Heart Failure (CHF), defined by:
* Presence of ≥2 of the following clinical signs and symptoms of congestion: jugular venous distension, pitting edema in lower extremities greater than trace, dyspnea, rales heard on auscultation, radiographic pulmonary congestion, weight gain above historical dry weight of at least 5 pounds (lbs) (2.27 Kilograms (kg)).
* Requiring treatment with intravenous (IV) diuretics.
* Estimated glomerular filtration rate (eGFR) ≥30 milliliter per minute (mL/min)/1.73 square meter (m^2) at the screening or randomization visit by the 4 variable Modification of Diet in Renal Disease (MDRD) equation.
* Female participants must use a double contraception method during the study including a highly effective method of birth control, except if she has undergone sterilization at least 3 months earlier or is postmenopausal.
* Male participants, unless vasectomized and confirmed sterile by sperm analysis, must use condoms during the study and refrain from donating sperm up to 90 days after the day of last dose. If the participant has a female partner of childbearing potential, the participant must wear a condom and female partner must use at least 1 highly effective method of birth control during the study treatment period and the Follow-up period.
* Transitioning from IV to oral diuretics, and oral diuretic treatment has been prescribed or administered.
* Hemodynamically stable, defined as systolic blood pressure (SBP) >100 millimeters of mercury (mmHg) with no requirement for IV inotropes or IV vasodilators.

Exclusion criteria :

* History of Type 1 diabetes mellitus.
* Appears unlikely or unable to participate in the required study procedures, as assessed by the study Investigator, study coordinator, or designee (ex: clinically-significant psychiatric, addictive, or neurological disease), or sectioned due to an official or court order.
* Current admission or visit for Worsening Heart Failure (HF) that is clearly and primarily triggered by causes such as tachyarrhythmia (example: sustained ventricular tachycardia, or atrial fibrillation/flutter with sustained ventricular response > 130 beats per minute), acute coronary syndrome, pulmonary embolism, cerebrovascular accident, heart valve disorders (such as severe aortic stenosis), as determined by the Investigator.
* Clinically significant myocardial infarction (MI) within past 1 month as determined by Investigator and with objective evidence from ECG, and/or cardiac imaging and/or coronary angiography. Small isolated elevations in troponin that often accompany HF hospitalization are not an exclusion, nor are clinically significant MIs that have been revascularized without complications.
* Participants who recently had or scheduled to have cardiac interventions may be eligible if:
* Stable 48 hours post procedure.
* Have diuretic treatment planned for the duration of treatment in this study.
* Current use of or recent suspension of digoxin therapy with high levels of digoxin (level should be obtained and must be <1.2 nanograms per milliliter (ng/mL) at screening.
* History of heart or kidney transplant.
* Diagnosis of hypertrophic obstructive cardiomyopathy.
* End-stage HF defined as requiring left ventricular assist device insertion, intra-aortic balloon placement (IABP), or any type of mechanical support during the study period.
* Pregnancy (demonstrated by serum pregnancy test at screening), breast-feeding, or inability or refusal to undergo pregnancy testing.
* Use of any investigational drug(s) or prohibited therapy or sodium-glucose co-transporter 2 (SGLT2) 5 half-lives prior to screening.
* Participants with moderate or severe respiratory, hepatic, neurological, psychiatric, active malignant tumor or other major systemic disease (including any diseases with evidence of malabsorption), making implementation of the protocol and/or the interpretation of the study results difficult.
* Known allergies, hypersensitivity, or intolerance to sotagliflozin or any inactive component of sotagliflozin or placebo (ie, microcrystalline cellulose, croscarmellose sodium [disintegrant], talc, silicon dioxide, and magnesium stearate [non-bovine]), unless the reaction is deemed irrelevant to the study by the PI.
* Laboratory findings at the Screening Visit:
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the upper limit of the normal laboratory range (ULN) (1 repeat lab allowed).
* Total bilirubin >1.7 times the ULN (except in case of Gilbert's syndrome) (1 repeat lab allowed).
* Amylase and/or lipase >3 times the ULN (1 repeat lab allowed).
* Participants with a severe or persistent in spite of optimal treatment genitourinary tract infection at time of randomization.
* Participant is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* History of diabetic ketoacidosis or non-ketotic hyperosmolar coma within 3 months prior to the screening visit.
* Lower extremity diabetic complications (such as skin ulcers, infection, osteomyelitis and gangrene) identified during the Screening period, and still requiring treatment at randomization.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-08-17 (Actual); Study Completion 2019-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (6):
- United States (4):
  - Investigational Site Number 8400005, La Jolla, California
  - Investigational Site Number 8400001, New Haven, Connecticut
  - Investigational Site Number 8400007, Rochester, Minnesota
  - Investigational Site Number 8400002, Cleveland, Ohio
- Investigational Site Number 1240001, Toronto, Canada
- Investigational Site Number 5280001, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the United States, Canada, and the Netherlands from 04 December 2017 to 17 August 2019.
Pre-assignment Details: Participants with a diagnosis of Congestive Heart Failure (CHF), were enrolled in 1 of 3 treatment groups: Placebo, Sotagliflozin 200 milligrams (mg) or Sotagliflozin 400 mg.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Started | 11 | 10 | 11
Completed | 10 | 10 | 10
Not Completed | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Did not Receive Treatment | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who had exposure to any amount of Investigational Medicinal Product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 10 | 10 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (13.05) | 55.1 (12.84) | 65.1 (13.41) | 60.5 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 4 | 7
  Male | 7 | 10 | 7 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 10 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 4 | 15
  White | 4 | 5 | 6 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Albumin [Mean (Standard Deviation); unit: gram per liter (g/L)] — Population: Pharmacodynamic (PD) population included all randomized and treated participants who had valid values of the main PD parameters at baseline.
  gram per liter (g/L)
    number analyzed (Participants) | 7 | 7 | 9 | 23
    (all) | 40.9 (3.48) | 38.0 (6.76) | 41.2 (2.59) | 40.1 (4.51)
Hematocrit [Mean (Standard Deviation); unit: percentage of red blood cells] — Population: PD population included all randomized and treated participants who had valid values of the main PD parameters at baseline.
  percentage of red blood cells
    number analyzed (Participants) | 10 | 10 | 10 | 30
    (all) | 0.38 (0.060) | 0.42 (0.092) | 0.39 (0.052) | 0.40 (0.070)
Hemoglobin [Mean (Standard Deviation); unit: g/L] — Population: PD population included all randomized and treated participants who had valid values of the main PD parameters at baseline.
  g/L
    number analyzed (Participants) | 10 | 10 | 10 | 30
    (all) | 119.6 (22.86) | 138.9 (28.23) | 124.4 (22.05) | 127.6 (25.10)
Total Protein [Mean (Standard Deviation); unit: g/L] — Population: PD population included all randomized and treated participants who had valid values of the main PD parameters at baseline.
  g/L
    number analyzed (Participants) | 7 | 7 | 9 | 23
    (all) | 69.0 (6.14) | 65.3 (9.88) | 69.6 (6.23) | 68.1 (7.39)
Plasma Volume [Mean (Standard Deviation); unit: milliliter (mL)] — Population: PD population included all randomized and treated participants who had valid values of the main PD parameters at baseline.
  milliliter (mL)
    number analyzed (Participants) | 4 | 6 | 6 | 16
    (all) | 3797.3 (1281.16) | 4489.3 (1306.41) | 3604.7 (1100.69) | 3984.6 (1212.44)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), AEs of Special Interest (AESIs), AEs Leading to Discontinuation From the Investigational Medicinal Product (IMP) and Deaths
Description: AE: is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. SAEs: an event that results in death; an event that, in the view of the investigator, places the participants at immediate risk of death (a life-threatening event); an outcome that results in a congenital anomaly/birth defect diagnosed in a child of a participant; an event that requires or prolongs inpatient hospitalization; an event that results in persistent or significant disability/incapacity. AESI: is an adverse event (serious or nonserious) of scientific and medical concern, specific to the IMP or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor may be appropriate.
Time Frame: Baseline up to Day 14
Population: Safety population included all randomized participants who had exposure to any amount of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 10 | 10 | 11
percentage of participants
  AEs | 40 | 30 | 45.5
  SAEs | 10 | 0 | 0
  AESIs | 0 | 0 | 0
  AEs Leading to Discontinuation From the IMP | 0 | 0 | 9.1
  Deaths | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Hemoconcentration as Assessed by Changes in Albumin to Day 14
Time Frame: Baseline to Day 14
Population: Pharmacodynamic (PD) population included all randomized and treated participants who had valid values of the main PD parameters at baseline and Day 14 End of Treatment (EOT). The number of participants analyzed is the number of participants with available data.
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 7 | 6 | 9
g/L | 1.17 (2.71) | 2.44 (2.40) | 0.15 (2.14)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; Analysis of Covariance (ANCOVA) model with fixed effects for treatment and stratification factors of baseline participant status (diabetic/non-diabetic, ejection fraction status (reduced/preserved) with baseline plasma volume as the covariate; Test type: Superiority; p = 0.736, ANCOVA; Difference in Least Squares (LS) Means = 1.26, 90% CI 2-sided [-5.4 to 7.93], Standard Error of Mean 3.64
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; ANCOVA model with fixed effects for treatment and stratification factors of baseline participant status (diabetic/non-diabetic, ejection fraction status (reduced/preserved) with baseline plasma volume as the covariate; Test type: Superiority; p = 0.7694, ANCOVA; Difference in LS Means = -1.02, 90% CI 2-sided [-7.22 to 5.18], Standard Error of Mean 3.38

3. Primary Outcome: Change From Baseline in Hemoconcentration as Assessed by Changes in Hematocrit to Day 14
Time Frame: Baseline to Day 14
Population: PD population included all randomized and treated participants who had valid values of the main PD parameters at baseline and Day 14 (EOT). The number of participants analyzed is the number of participants with available data.
Measure: Least Squares Mean (Standard Error); unit: percentage of red blood cells
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 10 | 9 | 10
percentage of red blood cells | 0.02 (0.02) | -0.02 (0.02) | -0.01 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; ANCOVA model with fixed effects for treatment and stratification factors of baseline participant status (diabetic/non-diabetic), ejection fraction status (reduced/preserved) with baseline plasma volume as the covariate; Test type: Superiority; p = 0.184, ANCOVA; Difference in LS Means = -0.04, 90% CI 2-sided [-0.09 to 0.01], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3397, ANCOVA; Difference in LS Means = -0.03, 90% CI 2-sided [-0.07 to 0.02], Standard Error of Mean 0.03

4. Primary Outcome: Change From Baseline in Hemoconcentration as Assessed by Changes in Hemoglobin to Day 14
Time Frame: Baseline to Day 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 10 | 9 | 10
g/L | 8.16 (6.80) | -8.91 (6.02) | -3.94 (5.37)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.094, ANCOVA; Difference in LS Means = -17.07, 90% CI 2-sided [-33.79 to -0.35], Standard Error of Mean 9.12
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1878, ANCOVA; Difference in LS Means = -12.09, 90% CI 2-sided [-27.65 to 3.46], Standard Error of Mean 8.49

5. Primary Outcome: Change From Baseline in Hemoconcentration as Assessed by Changes in Total Protein to Day 14
Time Frame: Baseline to Day 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 7 | 6 | 9
g/L | 5.31 (4.32) | 0.49 (3.83) | -1.05 (3.41)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4269, ANCOVA; Difference in LS Means = -4.82, 90% CI 2-sided [-15.45 to 5.8], Standard Error of Mean 5.8
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.2684, ANCOVA; Difference in LS Means = -6.36, 90% CI 2-sided [-16.24 to 3.52], Standard Error of Mean 5.39

6. Primary Outcome: Changes From Baseline in Plasma Volume to Day 14
Description: Change in plasma volume in milliliters (mL) was assessed by the indicator dilution method using 131I-labelled human albumin.
Time Frame: Baseline to 14 Days
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 4 | 6 | 5
mL | -525.00 (433.19) | 322.20 (359.23) | -35.67 (392.43)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1761, ANCOVA; Difference in LS Means = 847.2, 90% CI 2-sided [-210.46 to 1904.86], Standard Error of Mean 576.98
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4202, ANCOVA; Difference in LS Means = 489.33, 90% CI 2-sided [-572.68 to 1551.34], Standard Error of Mean 579.35

7. Secondary Outcome: Change From Baseline in Erythropoietin to Day 14
Description: Change in erythropoietin international units per liter (IU/L) was measured by chemiluminescent enzyme-labelled immunometric assay.
Time Frame: Baseline to Day 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 7 | 7 | 10
IU/L | 0.03 (5.92) | 13.78 (6.26) | -0.07 (5.04)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; ANCOVA model with fixed effects for treatment and stratification factors of baseline participant status (diabetic/non-diabetic), ejection fraction status (reduced/preserved) with baseline erythropoietin as the covariate; Test type: Superiority; p = 0.1242, ANCOVA; Difference in LS Means = 13.75, 90% CI 2-sided [-1.03 to 28.53], Standard Error of Mean 8.53
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.9903, ANCOVA; Difference in LS Means = 0.1, 90% CI 2-sided [-13.49 to 13.30], Standard Error of Mean 7.73

8. Secondary Outcome: Change From Baseline in N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP) to Day 14
Description: Change in NT-proBNP picomoles per liter (pmol/L) was measured by standard electrochemiluminescence immunoassay.
Time Frame: Baseline to Day 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 7 | 6 | 9
pmol/L | 91.36 (78.04) | -59.53 (81.28) | 86.10 (65.87)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; ANCOVA model with fixed effects for treatment and stratification factors of baseline participant status (diabetic/non-diabetic), ejection fraction status (reduced/preserved) with baseline NT-proBNP as the covariate; Test type: Superiority; p = 0.2121, ANCOVA; Difference in LS Means = -150.89, 90% CI 2-sided [-353.57 to 51.78], Standard Error of Mean 116.09
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.9574, ANCOVA; Difference in LS Means = -5.26, 90% CI 2-sided [-174.4 to 163.87], Standard Error of Mean 96.88

ADVERSE EVENTS:
Time Frame: First dose of study drug to last dose of study drug (up to Day 14) + 2 weeks
Description: Safety population included all randomized participants who had exposure to any amount of IMP.
Groups:
- Sotagliflozin 200 mg: Participants were randomized to Sotagliflozin 200 mg tablet administered as 1 sotagliflozin tablet and 1 matching placebo tablet, once daily, before the first meal of the day in the double-blind treatment period for up to 14 days.
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Sotagliflozin 200 mg (N=10) | Sotagliflozin 400 mg (N=11)
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Sotagliflozin 200 mg (N=10) | Sotagliflozin 400 mg (N=11)
Hypotension (Vascular disorders) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Fluid intake reduced (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT03292653/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT03292653/SAP_001.pdf